CLINICAL TRIAL: NCT04756232
Title: Cholinergic Mechanisms of Attention in Aging
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly Albert, Research Instructor, Psychiatry, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 210003
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Subjective Cognitive Decline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anticholinergic Challenge (Experimental): All participants will receive oral mecamylamine or IV scopolamine for 1 day
  Interventions: Drug: Mecamylamine Challenge
- Placebo Challenge (Placebo Comparator): All participants will receive oral placebo for 1 day
  Interventions: Other: Placebo Comparator Challenge

INTERVENTIONS:
Drug: Mecamylamine Challenge — Mecamylamine 20 mg oral pill administered once
  Arms: Anticholinergic Challenge
Other: Placebo Comparator Challenge — Matching placebo oral pill administered once
  Arms: Placebo Challenge

SUMMARY:
This study will use an anticholinergic pharmacological probe to examine attention network function in SCD using EEG. The overall hypothesis is that in older adults with SCD, normal cognitive performance is maintained by compensatory attention network activity, supported by enhanced cholinergic function. The investigators anticipate that SCD will be associated with greater compensatory attention network activity and that disrupting this compensatory process through anticholinergic challenge will result in a greater negative effect on attentional performance (Attention Network Test, ANT) and attention network functioning (EEG) in older adults with SCD compared to those without SCD.

DETAILED DESCRIPTION:
Overview: Cognitively normal older adults with and without subjective cognitive decline (SCD) (n = 20; SCD = 10, Non-SCD = 10) will complete two study visits that will be double blinded and randomized for anticholinergic challenge (mecamylamine/scopolamine or placebo). Drug challenge visits will include cognitive testing and an electroencephalography (EEG) session.

Aim 1: Feasibility of EEG during mecamylamine/scopolamine challenge

The primary outcome measures for Aim 1 will be the rate of completion of study visits with drug challenge and of completion of EEG tasks during the study visits with drug challenge.

Attention Network Test: The attention network test (ANT) is designed to test selective attention , and combines attentional cues with a flanker task. Behavioral measures of the ANT will be 1) Alerting: reaction time (RT) non-cue trials - cue trials; 2) Orienting: RT neutral cue trials - spatial cue trials; 3) Executive: RT incongruent trials - congruent trials.

EEG, Task-related Event Related Potentials: Each participant will complete the ANT during EEG with primary event relation potential (ERP) measures: 1) Alerting: early sensory ERP (P1) amplitude; 2) Orienting: early sensory ERP (P1) amplitude; 3) Executive: target and conflict evaluation ERP (P3) amplitude. Other ERP signals related to attention and sensory processing will be examined in exploratory analyses.

Incidental Memory: Incidental Memory Task during EEG, a passive visual memory paradigm that will allow an exploratory examination of the relationship between SCD and brain activity for memory recognition.

Psychomotor Speed: The Choice Reaction Time task will be used as a test of psychomotor speed. This task decomposes overall reaction time into recognition and motor components, allowing for the assessment of response and motor time that cannot be attained during the ANT.

Episodic Memory: The Selective Reminding Task (SRT) is a multi-trial verbal list-learning task that offers measures of storage into and retrieval from both short term and long term memory and intrusion errors. Outcome measures will be total recall (8 trials), total recall failures (8 trials), and delayed recall (20 minutes).

Study Drug Administration: During challenge drug study visits, participants will receive double-blinded administration of study drug (either 20 mg oral mecamylamine or 2.5 μg/kg intravenous scopolamine) or placebo. The order of administration will be randomized across study days. Randomization and dispensing will be managed by VUMC Investigational Drug Services.

Mecamylamine is a centrally and peripherally active non-competitive antagonist of nicotine (and presumably acetylcholine) at C6 (ganglionic) type nicotinic receptors. Peak cognitive and physiologic effects occur by 2-3 hours and dissipate by 4-6 hours after oral administration. Scopolamine is a centrally active antimuscarinic anticholinergic compound and is a competitive antagonist of the effects of acetylcholine on postganglionic cholinergic nerves. At the doses to be used in this study, the expected physiologic effects of scopolamine include cycloplegia, mydriasis, drowsiness, partial amnesia, decreased bowel motility, tachycardia and decreased salivation. After intravenous administration, the early effects of scopolamine include tachycardia, dryness of mouth, and inhibition of lacrimation and sweating. Memory and attention changes are maximal between 90 and l50 minutes after an IV dose. The drug is distributed throughout the body with a serum half-life of approximately 2-3 hours. We have used both mecamylamine and scopolamine extensively in clinical studies in identical doses to those proposed here.

Statistical Analysis Plan:This project is a pilot study to determine the feasibility and participant tolerability for conducting EEG during the mecamylamine/scopolamine challenge. The proposed sample size (n =20) is designed to provide sufficient experience with the protocol to determine our ability to complete this protocol in a larger study and determine completion rates for the two participant groups (SCD and Non-SCD) as preliminary data for an NIH K01 application resubmission for Dr. Albert. Dr. Hakmook Kang is the biostatistics consultant for this project.

Descriptive statistics will be used to identify the rate of completion of study visits with drug challenge (proportion of participants that complete both study days), and of completion of EEG tasks (proportion of participants who complete both tasks on each study visits with drug challenge). These measures will be calculated for all participants (n = 20), and for participant groups separately (SCD, n = 10; Non-SCD, n = 10).

The investigators have hypothesized that > 80 % of participants will complete both study visits with drug challenge based on their experience using anticholinergic challenge with 88% of participants completing 2 study visits including anticholinergic challengeor placebo administration. The investigators have hypothesized that > 70 % of participants will complete both EEG tasks (ANT and incidental memory) during study visits with drug challenge, based on previous completion rates of 72% for non-EEG tasks during study visits including anticholinergic challenge or placebo administration, and 100% for EEG tasks with no drug challenge.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 55
2. Montreal Cognitive Assessment (MoCA) > 25 AND Global Deterioration Scale (GDS) rating < 3
3. Non-smokers

Exclusion Criteria:

1. medical contraindications to the drug challenge
2. primary neurological disorder (such as stroke, epilepsy, etc.)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who complete study visits with drug challenge | After administration of second drug challenge, approximately 72 hours
  Proportion of particiapnts who complete study days as measured by study drug administration on both study visits with drug challenge
Proportion of participants who complete EEG | After administration of second drug challenge, approximately 72 hours
  Proportion of participants who complete EEG sessions as measured by adminstration of EEG

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newhouse, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No